CLINICAL TRIAL: NCT04727385
Title: First-in-human Pilot Study for the Safety Assessment of DXM Gel in Patients With Painful Lumbar Degenerative Disc Disease
Brief Title: Intervertebral DXM Gel Injection in Adults With Painful Lumbar Degenerative Disc Disease
Acronym: DXM gel
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gelmetix (Industry)
Collaborators: Excelya (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-A02476-51
Record Dates: First submitted 2021-01-13; First posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Degenerative Disc Disease; Chronic Lower Back Pain; Discogenic Pain; Intervertebral Disc Degeneration; Lumbar Disc Disease; Lumbar Disc Degeneration; Lumbar Disc Pain
Keywords: Degenerative Disc Disease; Chronic Lower Back Pain; Double Cross-Linked hydrogel; disc nucleus; medical device; Double Crosslink Microgel; first in human; intervertebral disc space; Oswestry Disability Index; discs partial dehydration; proteoglycan matrix; Pfirrmann classification; inter-vertebral disc water content
MeSH Terms: conditions — Intervertebral Disc Degeneration; Intervertebral disc disease

STUDY DESIGN:
Intervention Model Description: This is an adaptative-design, interventional, open-label, single-arm trial performed at a single centre in France.
  3 cohorts will be sequentially initiated according to the DSMB review of the safety parameters :
  The safety primary endpoints of each cohort will be assessed by an independent Data Safety Monitoring Board (DSMB) at Day 42 post-injection to provide safety oversight on the patients and guidance on initiating the study on the next cohort.
  Patients will be injected at day 0 and will be followed-up for a variable period according to the cohort.
  * As the first enrolled cohort, the 1L cohort will have the longest follow-up (48 weeks) and will attend 9 visits.
  * The second cohort (2L) will have a shorter follow-up period (36 weeks) attend the same visits except for V9, which will not be done.
  * The third cohort (1-2L) will will have the shorter follow-up period (24 weeks) and will attend visits 1 to 7 except for V4, which will not be done.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single-arm of 3 cohorts (Experimental): These patients will be sequentially recruited in 3 cohorts :
  * One disc level cohort: 5 patients with only one disc to be treated; First enrolled cohort with 48 weeks of follow-up (9 visits V1-V9)
  * Two disc level cohort: 5 patients with 2 discs to be treated; Second enrolled cohort with 36 weeks of follow-up (8 visits, same visits except for V9)
  * One or two disc level cohort: 10 patients with 1 or 2 discs to be treated; Third enrolled cohort with 24 weeks of follow-up (6 visits, V1 to 7 except for V4)
  Interventions: Device: Double Crosslink Microgel

INTERVENTIONS:
Device: Double Crosslink Microgel — DXM hydrogel is a pH responsive Double Cross-Linked microgel based on single internally cross-linked microspheres (comprising a methacrylic acid-methyl methacrylate-ethylene glycol dimethacrylate copolymer)
  The DXM gel is injected into the intervertebral disc (IVD) space via a standardised procedure similar to the routinely-performed Discography procedure. The disc approach described in the discography procedure has been reported to allow the injection of a solution in the centre of the disc. The injection of the gel takes about 2 min.
  Other Names: DXM gel

SUMMARY:
The purpose of this study is to assess the safety and the efficacy of an hydrogel (double cross-link microgel - DXM) injection into the intervertebral disc (IVD) space in patients with painful lumbar degenerative disc disease (DDD) over 24 to 48 weeks.

DETAILED DESCRIPTION:
After being informed of the study and the potential risks, all patients matching the eligibility criteria and who have given their written consent will undergo a gel injection at day 0 after a period of screening of up to 14 days.

Then, they will be followed-up for a variable period according to the cohort :

* first cohort of 5 patients with only one disc to be treated will be followed during 48 weeks,
* second cohort of 5 patients with 2 discs to be treated will be followed during 36 weeks,
* third cohort of 10 patients with 1 or 2 discs to be treated will be followed during 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient aged between 18 and 55 (inclusive)
2. Discogenic low back pain, confirmed by a history of Low Back Pain, with a minimum of 3 months of continuous pain or 6 months of acute episodes of pain despite the conservative treatment including painkillers and physiotherapy
3. Oswestry Disability Index (ODI) ≥ 30% and ≤ 60%,
4. Painful disc(s) between L1 and S1 represented

   1. For cohort 1L: at a single disc level
   2. For cohort 2L: at 2 disc levels
   3. For cohort 1-2L: at 1 or 2 disc levels
5. Patients with a Zung depression score ≤ 49, Note: Patients with a Zung depression score between ≥ 50 and ≤ 64 may be included if deemed suitable for trial inclusion by the investigator
6. Partial dehydration (grey disc) confirmed by MRI, grade II/III Pfirrmann classification

   Note:
   * Pfirrmann Grade I lesions are not contra-indications to recruitment, but can never be the target of any intervention in this trial. Patients featuring grade I disc(s) in conjunction with a grade II/III meet the inclusion criteria for his(her) disc Grade II/III disc to be treated
   * Pfirrmann Grade IV and V disc lesions are absolute contra-indications for inclusion
7. Female patients of childbearing potential must have a negative urine pregnancy test at screening and use an effective birth control during the follow up period after the injection procedure
8. Patients who are willing and capable of understanding the investigator's explanations, following his instructions and adhering to the follow-up visits according to the study protocol, including a willingness and ability to undergo MRI scanning,
9. Patient giving informed consent to take part in the study

Exclusion Criteria:

1. Averted nerve root pain and potential root compression Note: Referred leg pain authorised
2. Presence of posterior bone spurs (osteophytes)
3. Partial or total Modic signal grade 1 at the considered disc level
4. Patients with active systemic infection or infection localized to the site of the proposed implantation.
5. Any conditions not described in the indications for use.
6. Any mental conditions or neuromuscular disease that may generate an unacceptable risk of failure or postoperative complication.
7. Patients with existing disc herniation at the considered level and on adjacent discs
8. Endplate disease, defect or weakness, e.g. Schmorl nodule
9. Vertebral bone abnormalities with active angioma
10. Disc collapse ≥ 15% when disc height is compared to the height of the upper adjacent disc
11. One lumbar disc rated grade IV or V on the Pfirrmann classification
12. Imaging showing facet arthrosis
13. Lytic spondylolisthesis
14. Degenerative spondylolisthesis grade > grade I Meyerding
15. Congenital or idiopathic deformities of the spine (e.g. Scoliosis >20° Cobb or Kyphosis)
16. Old or acute vertebral fractures in the lumbar spine
17. Patients with any prior spine procedure in the lumbar spine
18. Any skin disease or inadequate tissue coverage at the site of the injection
19. Any medical or surgical conditions that could preclude the potential benefit of disc injection must be carefully analysed before the procedure, such as congenital abnormalities, immunosuppressive disease, elevation of erythrocyte sedimentation rate (ESR) or C-reactive protein (CRP) concentration not explained by other diseases, elevation of white blood cell (WBC) count, or marked left shift in the WBC differential count, should be carefully taken into consideration prior to the surgical procedure.

    Note: These contra-indications can be relative or absolute and must be taken into account by the physician when making his decision. The above list is not exhaustive.
20. Tumours with any metastatic potential, or known metastases, in any part of the body
21. Known infection with HIV or Hepatitis B, C or E
22. Patient that has received or is seeking employee compensation
23. Zung depression score ≥ 65
24. Substance abuse or dependency (pharmaceuticals, drugs, alcohol)
25. Disabling obesity (BMI > 35kg/m²)
26. History of chemical dependency (e.g. illicit drugs, or opiates) or significant emotional or psychosocial disturbance which may have an effect on treatment outcome
27. Patients who are pregnant, breast feeding or planning pregnancy during the study
28. Anticoagulation (beyond low level prophylactic doses of single anti-platelet agents)
29. Inability to undertake or known contra-indications to MRI scanning
30. Known hypersensitivity to barium sulphate

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
The number of patients with at least one adverse event (AE) or serious adverse event (SAE) | Between screening visit and 24 weeks (measured at each visits)
  An adverse event (AE) is any untoward medical occurrence in a patient exposed to a medical device and which does not necessarily have a causal relationship with this medical device.
  An AE can therefore be any unintended disease or injury or clinical signs (including an abnormal laboratory finding) in subjects, users or other persons whether or not considered related to the investigational medical device.
  A serious adverse event (SAE) is defined as an AE that:
  * led to a death, injury or permanent impairment to a body structure or a body function;
  * led to a serious deterioration in health of the subject, that either resulted in: a life-threatening illness or injury, or a permanent impairment of a body structure or a body function, or in-patient hospitalization or prolongation of existing hospitalization, or in medical or surgical intervention to prevent life threatening illness
  * led to foetal distress, foetal death or a congenital abnormality or birth defect.
The number of adverse events (AEs) or serious adverse event (SAEs) | Between screening visit and 24 weeks (measured at each visits)
  An adverse event (AE) is any untoward medical occurrence in a patient exposed to a medical device and which does not necessarily have a causal relationship with this medical device.
  An AE can therefore be any unintended disease or injury or clinical signs (including an abnormal laboratory finding) in subjects, users or other persons whether or not considered related to the investigational medical device.
  A serious adverse event (SAE) is defined as an AE that:
  * led to a death, injury or permanent impairment to a body structure or a body function;
  * led to a serious deterioration in health of the subject, that either resulted in: a life-threatening illness or injury, or a permanent impairment of a body structure or a body function, or in-patient hospitalization or prolongation of existing hospitalization, or in medical or surgical intervention to prevent life threatening illness
  * led to foetal distress, foetal death or a congenital abnormality or birth defect.
The number of patients with neurological changes during the follow-up period according to the evaluation of nerve root pain, sensory deficit and motor deficit | Between screening visit and 24 weeks (measured at each visits)
  The neurological evaluation will look more specifically for:
  * The presence or absence of nerve root pain and its localisation (i.e. Lassegue test)
  * The presence of deferred pain in the leg without deficit
  * The presence or absence of sensory deficit and its localisation
  * The presence or absence of motor deficit and its classification from grade 1 to 5 (0 - Total Paralysis, 1 - Palpable or Visible, 2 - Active Movement, gravity eliminated, 3 - Active Movement, against gravity, Contraction, 4 - Active Movement, against some resistance, 5 - Active Movement, against full resistance (normal muscular force))
The change of the water content of the nucleus measured in milliseconds on the MRI during the follow-up period | Between screening visit and 24 weeks (measured at each visits)
  The Magnetic resonance imaging (MRI) will allow the observation.
The modifications observed after the injection in the adjacent tissues of the injected nucleus | Between screening visit and 24 weeks (measured at each visits)
  The Magnetic resonance imaging (MRI) will allow the observation of the corresponding adjacent tissues:
  * Annulus fibrosus
  * Endplates
  * Facets
The change of the intervertebral height in millimetres of the injected disc | Between screening visit and 24 weeks (measured at each visits)
  The Magnetic resonance imaging (MRI) will allow the observation.
The change of the DXM gel position in relation to posterior and anterior limit of the annulus fibrosus and vertebral disc end-plates | Between screening visit and 24 weeks (measured at each visits)
  The Magnetic resonance imaging (MRI) will allow the observation.

SECONDARY OUTCOMES:
The number of patients with at least one adverse event (AE) or serious adverse event (SAE) | Over 48 weeks for the first cohort (1L) / 36 weeks for the second cohort (2L) / 24 weeks for the third cohort (1-2L)
  An adverse event (AE) is any untoward medical occurrence in a patient exposed to a medical device and which does not necessarily have a causal relationship with this medical device.
  An AE can therefore be any unintended disease or injury or clinical signs (including an abnormal laboratory finding) in subjects, users or other persons whether or not considered related to the investigational medical device.
  A serious adverse event (SAE) is defined as an AE that:
  * led to a death, injury or permanent impairment to a body structure or a body function;
  * led to a serious deterioration in health of the subject, that either resulted in: a life-threatening illness or injury, or a permanent impairment of a body structure or a body function, or in-patient hospitalization or prolongation of existing hospitalization, or in medical or surgical intervention to prevent life threatening illness
  * led to foetal distress, foetal death or a congenital abnormality or birth defect.
The number of adverse events (AEs) or serious adverse event (SAEs) | Over 48 weeks for the first cohort (1L) / 36 weeks for the second cohort (2L) / 24 weeks for the third cohort (1-2L)
  An adverse event (AE) is any untoward medical occurrence in a patient exposed to a medical device and which does not necessarily have a causal relationship with this medical device.
  An AE can therefore be any unintended disease or injury or clinical signs (including an abnormal laboratory finding) in subjects, users or other persons whether or not considered related to the investigational medical device.
  A serious adverse event (SAE) is defined as an AE that:
  * led to a death, injury or permanent impairment to a body structure or a body function;
  * led to a serious deterioration in health of the subject, that either resulted in: a life-threatening illness or injury, or a permanent impairment of a body structure or a body function, or in-patient hospitalization or prolongation of existing hospitalization, or in medical or surgical intervention to prevent life threatening illness
  * led to foetal distress, foetal death or a congenital abnormality or birth defect.
The number of patients with neurological changes during the follow-up period according to the evaluation of nerve root pain, sensory deficit and motor deficit | Over 48 weeks for the first cohort (1L) / 36 weeks for the second cohort (2L) / 24 weeks for the third cohort (1-2L)
  The neurological evaluation will look more specifically for:
  * The presence or absence of nerve root pain and its localisation (i.e. Lassegue test)
  * The presence of deferred pain in the leg without deficit
  * The presence or absence of sensory deficit and its localisation
  * The presence or absence of motor deficit and its classification from grade 1 to 5 (0 - Total Paralysis, 1 - Palpable or Visible, 2 - Active Movement, gravity eliminated, 3 - Active Movement, against gravity, Contraction, 4 - Active Movement, against some resistance, 5 - Active Movement, against full resistance (normal muscular force))
The change of the water content of the nucleus measured in milliseconds on the MRI during the follow-up period | Over 48 weeks for the first cohort (1L) / 36 weeks for the second cohort (2L) / 24 weeks for the third cohort (1-2L)
  The Magnetic resonance imaging (MRI) will allow the observation.
The modifications observed after the injection in the adjacent tissues of the injected nucleus | Over 48 weeks for the first cohort (1L) / 36 weeks for the second cohort (2L) / 24 weeks for the third cohort (1-2L)
  The Magnetic resonance imaging (MRI) will allow the observation of the corresponding adjacent tissues:
  * Annulus fibrosus
  * Endplates
  * Facets
The change of the intervertebral height in millimetres of the injected disc | Over 48 weeks for the first cohort (1L) / 36 weeks for the second cohort (2L) / 24 weeks for the third cohort (1-2L)
  The Magnetic resonance imaging (MRI) will allow the observation.
The change of the DXM gel position in relation to posterior and anterior limit of the annulus fibrosus and vertebral disc end-plates | Over 48 weeks for the first cohort (1L) / 36 weeks for the second cohort (2L) / 24 weeks for the third cohort (1-2L)
  The Magnetic resonance imaging (MRI) will allow the observation.
Oswestry disability index (ODI) | Measured and compared to baseline at the different time points of the flowchart according to the cohort (over 24 to 48 weeks)
  The ODI score is based on a self-completed questionnaire of 10 items to measure a patient's permanent functional disability. It is a well-recognised, gold standard orthopaedic score devised in 1980 and which still remains the best and most reliable measure of the overall impact of spinal disease associated with low back pain and any interventions patients may receive. It has been repeatedly used for natural history studies, cohort studies, and for many device and surgery interventions. It is reproducible, reliable and responsive to therapeutic interventions.
Visual analogue scale (VAS) self-assessment | Measured and compared to baseline at the different time points of the flowchart according to the cohort (over 24 to 48 weeks)
  The visual analogue self-assessment scale is an evaluation performed by the patient to specify his level of pain on a scale of 'no pain' to 'extreme pain'.
  During the site visit, the VAS is to be filled on-site by the patient and collected by the site staff.
Working status | measured and compared to baseline at the different time points of the flowchart according to the cohort (over 24 to 48 weeks)
  The working status will be collected by interviewing the patient about his/her work activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Polyclinique Bordeaux Nord Aquitaine Centre Vertebra, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No